CLINICAL TRIAL: NCT00000608
Title: Dietary Patterns, Sodium Intake and Blood Pressure (DASH - Sodium)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Model: Parallel | Purpose: Prevention
Other Study IDs: 111; U01HL057139 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Fat-Restricted; Diet, Sodium-Restricted

INTERVENTIONS:
Behavioral: diet, fat-restricted
Behavioral: diet, sodium-restricted

SUMMARY:
To compare the effects of three levels of dietary sodium and two patterns of diet (a control diet and an intervention diet high in fruits, vegetables, and low fat dairy products and low in fat) on blood pressure in individuals with higher than optimal blood pressure or with Stage 1 hypertension.. DASH - Sodium built on and extended the results of the NHLBI-initiated Dietary Approaches to Stop Hypertension (DASH) study.

DETAILED DESCRIPTION:
BACKGROUND:

High blood pressure, defined as systolic blood pressure greater than or equal to 140 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg, or taking antihypertensive medication, affects 24 percent of the United States adult population or about 50 million people. Because the risk of cardiovascular disease and stroke increases with increasing blood pressure throughout the entire range of blood pressure levels, people with blood pressure above the optimal level of 120/80 are at increased risk of disease. Approximately 48 percent of the adult population have blood pressure either normal but above optimal levels or have Stage 1 hypertension, a prevalence which increases with age. To combat this highly prevalent condition, primary prevention through lifestyle modification represents a highly promising strategy for public health.

DASH - Sodium extended research from DASH trial to address several issues of relevance to clinical practice and public health and capitalized on the success of DASH by following the multicenter outpatient feeding study model. The model permitted a true test of efficacy because of high adherence and follow-up rates. In addition, the population studied across four geographic areas, encompassing individuals with diastolic blood pressure between 80-95 mm Hg and systolic blood pressure <160 mm Hg, was broadly representative, thus making the results generalizable to a large portion of the United States population.

DESIGN NARRATIVE:

The effects on blood pressure of three levels of sodium intake and two dietary patterns were compared. The combined impact of sodium reduction with dietary intervention was evaluated as a potential non-pharmacologic treatment alternative to drug therapy for stage one hypertension or for maintaining normal blood pressure levels. The two dietary patterns were a control diet that represented the typical American diet and an intervention diet (DASH diet) that was high in fruits, vegetables, included whole grains, poultry, fish, and nuts, and reduced in fats, red meat, sweets, and sugar-containing beverages and dairy products. The three levels of sodium were higher (current United States intake), intermediate (current recommended levels), and lower (potentially optimal levels). Participants were assigned to one of the two dietary patterns using a parallel group design and were fed at each sodium level using a randomized cross-over design.

Three eligibility pre-screening visits were followed by a two-week run-in feeding period and then a four-week intervention period at each of three sodium levels. During the run-in for the intervention feeding periods, all food was provided to participants. They were required to attend the clinic for at least one meal per day, five days per week, and to take home food to eat for other meals. Each of the four clinics recruited 100 participants. Blood pressure was measured once a week during the first of three weeks and five times during the last week. During the final feeding period, fasting blood was collected and 24-hour urine collections were analyzed for magnesium, potassium. calcium, sodium, and creatinine.

DASH - Sodium determined, separately by race, gender, and hypertension status: 1) the effects on blood pressure of three levels of dietary sodium within the context of both a control diet and the DASH diet; 2) the effect on blood pressure of the DASH diet, relative to the control diet, at each of the three levels of sodium intake. The study also assessed whether the effect on blood pressure of going from higher to lower sodium diets differs for participants in the control and DASH diets. Lastly, the study determined whether the blood pressure effect associated with reducing sodium from the higher to the intermediate level differs from the blood pressure effect associated with reducing sodium from the intermediate to the lower level, that is, testing whether the blood pressure effects of sodium are linear across sodium levels for each diet.

Recruitment and screening began in August 1997. The first cohort began the experimental diets in January 1998 and the last cohort completed the diets in November 1999. A total of 412 participants were enrolled into the study. Results were presented at the annual meeting of American Society of Hypertension in May 2000.

The study was renewed under R01HL57114 to to analyze the data of the trial The hypothesis to be tested is that genetic makeup modulates the BP effects of DASH diet and reduced sodium intake through one or more of the following mechanisms: 1) effects on vascular tone; 2) effects on mineralocorticoid regulation of sodium homeostasis; and 3) effects on non-classical regulation of sodium homeostasis.

ELIGIBILITY:
Healthy adult men and women, ages 22 and older, who had a diastolic blood pressure of 80 to 95 mm Hg and a systolic blood pressure less than 160 mm Hg.

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-02; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Vollmer — Kaiser Foundation Research Institute

REFERENCES:
- [Background] Svetkey LP, Sacks FM, Obarzanek E, Vollmer WM, Appel LJ, Lin PH, Karanja NM, Harsha DW, Bray GA, Aickin M, Proschan MA, Windhauser MM, Swain JF, McCarron PB, Rhodes DG, Laws RL. The DASH Diet, Sodium Intake and Blood Pressure Trial (DASH-sodium): rationale and design. DASH-Sodium Collaborative Research Group. J Am Diet Assoc. 1999 Aug;99(8 Suppl):S96-104. doi: 10.1016/s0002-8223(99)00423-x. PMID 10450301
- [Background] Greenland P. Beating high blood pressure with low-sodium DASH. N Engl J Med. 2001 Jan 4;344(1):53-5. doi: 10.1056/NEJM200101043440109. No abstract available. PMID 11136961
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Vollmer WM, Sacks FM, Ard J, Appel LJ, Bray GA, Simons-Morton DG, Conlin PR, Svetkey LP, Erlinger TP, Moore TJ, Karanja N; DASH-Sodium Trial Collaborative Research Group. Effects of diet and sodium intake on blood pressure: subgroup analysis of the DASH-sodium trial. Ann Intern Med. 2001 Dec 18;135(12):1019-28. doi: 10.7326/0003-4819-135-12-200112180-00005. PMID 11747380
- [Background] Phillips KM, Simpkins AH, Amanna KR, Wolf W, Stewart KK, Clark S, Kim KP, Beecher GR, Holden J. Long-term stability of nutrients in a frozen mixed food control material. Fresenius J Anal Chem. 2001 Jun;370(2-3):297-302. doi: 10.1007/s002160100785. PMID 11451255
- [Background] Conlin PR, Erlinger TP, Bohannon A, Miller ER 3rd, Appel LJ, Svetkey LP, Moore TJ. The DASH diet enhances the blood pressure response to losartan in hypertensive patients. Am J Hypertens. 2003 May;16(5 Pt 1):337-42. doi: 10.1016/s0895-7061(03)00056-6. PMID 12745193
- [Background] Lin PH, Aickin M, Champagne C, Craddick S, Sacks FM, McCarron P, Most-Windhauser MM, Rukenbrod F, Haworth L; Dash-Sodium Collaborative Research Group. Food group sources of nutrients in the dietary patterns of the DASH-Sodium trial. J Am Diet Assoc. 2003 Apr;103(4):488-96. doi: 10.1053/jada.2003.50065. PMID 12669013
- [Background] Erlinger TP, Miller ER 3rd, Charleston J, Appel LJ. Inflammation modifies the effects of a reduced-fat low-cholesterol diet on lipids: results from the DASH-sodium trial. Circulation. 2003 Jul 15;108(2):150-4. doi: 10.1161/01.CIR.0000080288.30567.86. Epub 2003 Jul 7. PMID 12847067
- [Background] Akita S, Sacks FM, Svetkey LP, Conlin PR, Kimura G; DASH-Sodium Trial Collaborative Research Group. Effects of the Dietary Approaches to Stop Hypertension (DASH) diet on the pressure-natriuresis relationship. Hypertension. 2003 Jul;42(1):8-13. doi: 10.1161/01.HYP.0000074668.08704.6E. Epub 2003 May 19. PMID 12756219
- [Background] Jurgens G, Graudal N; Dietary Approaches to Stop Hypertension. Subgroup results in the DASH-sodium trial. Ann Intern Med. 2002 Nov 5;137(9):772-3; author reply 772-3. doi: 10.7326/0003-4819-137-9-200211050-00018. No abstract available. PMID 12416957
- [Background] Harsha DW, Sacks FM, Obarzanek E, Svetkey LP, Lin PH, Bray GA, Aickin M, Conlin PR, Miller ER 3rd, Appel LJ. Effect of dietary sodium intake on blood lipids: results from the DASH-sodium trial. Hypertension. 2004 Feb;43(2):393-8. doi: 10.1161/01.HYP.0000113046.83819.a2. Epub 2004 Jan 5. PMID 14707154
- [Background] Most MM, Craddick S, Crawford S, Redican S, Rhodes D, Rukenbrod F, Laws R; Dash-Sodium Collaborative Research Group. Dietary quality assurance processes of the DASH-Sodium controlled diet study. J Am Diet Assoc. 2003 Oct;103(10):1339-46. doi: 10.1016/s0002-8223(03)01080-0. PMID 14520254
- [Background] Obarzanek E, Proschan MA, Vollmer WM, Moore TJ, Sacks FM, Appel LJ, Svetkey LP, Most-Windhauser MM, Cutler JA. Individual blood pressure responses to changes in salt intake: results from the DASH-Sodium trial. Hypertension. 2003 Oct;42(4):459-67. doi: 10.1161/01.HYP.0000091267.39066.72. Epub 2003 Sep 2. PMID 12953018
- [Background] Bray GA, Vollmer WM, Sacks FM, Obarzanek E, Svetkey LP, Appel LJ; DASH Collaborative Research Group. A further subgroup analysis of the effects of the DASH diet and three dietary sodium levels on blood pressure: results of the DASH-Sodium Trial. Am J Cardiol. 2004 Jul 15;94(2):222-7. doi: 10.1016/j.amjcard.2004.03.070. PMID 15246908
- [Background] Svetkey LP, Simons-Morton DG, Proschan MA, Sacks FM, Conlin PR, Harsha D, Moore TJ. Effect of the dietary approaches to stop hypertension diet and reduced sodium intake on blood pressure control. J Clin Hypertens (Greenwich). 2004 Jul;6(7):373-81. doi: 10.1111/j.1524-6175.2004.03523.x. PMID 15249792
- [Background] Ard JD, Coffman CJ, Lin PH, Svetkey LP. One-year follow-up study of blood pressure and dietary patterns in dietary approaches to stop hypertension (DASH)-sodium participants. Am J Hypertens. 2004 Dec;17(12 Pt 1):1156-62. doi: 10.1016/j.amjhyper.2004.07.005. PMID 15607623
- [Background] Kennedy BM, Conlin PR, Ernst D, Reams P, Charleston JB, Appel LJ. Successfully recruiting a multicultural population: the DASH-Sodium experience. Ethn Dis. 2005 Winter;15(1):123-9. PMID 15720059
- [Derived] Zheng X, Nist KM, Velkoska E, Wainford RD. Plasma and Urinary Metabolomic Profiles Associated with the Salt Sensitivity of Blood Pressure in the Dietary Approaches to Stop Hypertension-Sodium Trial. J Nutr. 2025 Nov 11:S0022-3166(25)00703-5. doi: 10.1016/j.tjnut.2025.11.007. Online ahead of print. PMID 41232772
- [Derived] Kim H, Lichtenstein AH, Coresh J, Appel LJ, Rebholz CM. Serum proteins associated with LDL-C and non-HDL-C reduction in response to dietary interventions in the DASH and DASH-Sodium trials. Food Funct. 2025 Nov 10;16(22):8764-8772. doi: 10.1039/d5fo02593a. PMID 41143495
- [Derived] Kim H, Appel LJ, Lichtenstein AH, Wong KE, Chatterjee N, Rhee EP, Rebholz CM. Metabolomic Profiles Associated With Blood Pressure Reduction in Response to the DASH and DASH-Sodium Dietary Interventions. Hypertension. 2023 Jul;80(7):1494-1506. doi: 10.1161/HYPERTENSIONAHA.123.20901. Epub 2023 May 10. PMID 37161796
- [Derived] Kim H, Lichtenstein AH, Ganz P, Du S, Tang O, Yu B, Chatterjee N, Appel LJ, Coresh J, Rebholz CM. Identification of Protein Biomarkers of the Dietary Approaches to Stop Hypertension Diet in Randomized Feeding Studies and Validation in an Observational Study. J Am Heart Assoc. 2023 Apr 4;12(7):e028821. doi: 10.1161/JAHA.122.028821. Epub 2023 Mar 28. PMID 36974735
- [Derived] Belanger MJ, Kovell LC, Turkson-Ocran RA, Mukamal KJ, Liu X, Appel LJ, Miller ER 3rd, Sacks FM, Christenson RH, Rebuck H, Chang AR, Juraschek SP. Effects of the Dietary Approaches to Stop Hypertension Diet on Change in Cardiac Biomarkers Over Time: Results From the DASH-Sodium Trial. J Am Heart Assoc. 2023 Jan 17;12(2):e026684. doi: 10.1161/JAHA.122.026684. Epub 2023 Jan 11. PMID 36628985
- [Derived] Juraschek SP, Kovell LC, Appel LJ, Miller ER 3rd, Sacks FM, Chang AR, Christenson RH, Rebuck H, Mukamal KJ. Effects of Diet and Sodium Reduction on Cardiac Injury, Strain, and Inflammation: The DASH-Sodium Trial. J Am Coll Cardiol. 2021 Jun 1;77(21):2625-2634. doi: 10.1016/j.jacc.2021.03.320. PMID 34045018
- [Derived] Chaudhary P, Velkoska E, Wainford RD. An exploratory analysis of comparative plasma metabolomic and lipidomic profiling in salt-sensitive and salt-resistant individuals from The Dietary Approaches to Stop Hypertension Sodium Trial. J Hypertens. 2021 Oct 1;39(10):1972-1981. doi: 10.1097/HJH.0000000000002904. PMID 34001808
- [Derived] Kim H, Lichtenstein AH, Wong KE, Appel LJ, Coresh J, Rebholz CM. Urine Metabolites Associated with the Dietary Approaches to Stop Hypertension (DASH) Diet: Results from the DASH-Sodium Trial. Mol Nutr Food Res. 2021 Feb;65(3):e2000695. doi: 10.1002/mnfr.202000695. Epub 2020 Dec 28. PMID 33300290
- [Derived] Juraschek SP, Miller ER 3rd, Chang AR, Anderson CAM, Hall JE, Appel LJ. Effects of Sodium Reduction on Energy, Metabolism, Weight, Thirst, and Urine Volume: Results From the DASH (Dietary Approaches to Stop Hypertension)-Sodium Trial. Hypertension. 2020 Mar;75(3):723-729. doi: 10.1161/HYPERTENSIONAHA.119.13932. Epub 2020 Jan 20. PMID 31957521
- [Derived] Peng AW, Juraschek SP, Appel LJ, Miller ER 3rd, Mueller NT. Effects of the DASH Diet and Sodium Intake on Bloating: Results From the DASH-Sodium Trial. Am J Gastroenterol. 2019 Jul;114(7):1109-1115. doi: 10.14309/ajg.0000000000000283. PMID 31206400
- [Derived] Peng AW, Appel LJ, Mueller NT, Tang O, Miller ER 3rd, Juraschek SP. Effects of sodium intake on postural lightheadedness: Results from the DASH-sodium trial. J Clin Hypertens (Greenwich). 2019 Mar;21(3):355-362. doi: 10.1111/jch.13487. Epub 2019 Jan 28. PMID 30690866
- [Derived] Juraschek SP, Miller ER 3rd, Weaver CM, Appel LJ. Effects of Sodium Reduction and the DASH Diet in Relation to Baseline Blood Pressure. J Am Coll Cardiol. 2017 Dec 12;70(23):2841-2848. doi: 10.1016/j.jacc.2017.10.011. Epub 2017 Nov 12. PMID 29141784
- [Derived] Juraschek SP, Woodward M, Sacks FM, Carey VJ, Miller ER 3rd, Appel LJ. Time Course of Change in Blood Pressure From Sodium Reduction and the DASH Diet. Hypertension. 2017 Nov;70(5):923-929. doi: 10.1161/HYPERTENSIONAHA.117.10017. PMID 28993451
- [Derived] Derkach A, Sampson J, Joseph J, Playdon MC, Stolzenberg-Solomon RZ. Effects of dietary sodium on metabolites: the Dietary Approaches to Stop Hypertension (DASH)-Sodium Feeding Study. Am J Clin Nutr. 2017 Oct;106(4):1131-1141. doi: 10.3945/ajcn.116.150136. Epub 2017 Aug 30. PMID 28855223
- [Derived] Juraschek SP, Choi HK, Tang O, Appel LJ, Miller ER 3rd. Opposing effects of sodium intake on uric acid and blood pressure and their causal implication. J Am Soc Hypertens. 2016 Dec;10(12):939-946.e2. doi: 10.1016/j.jash.2016.10.012. Epub 2016 Nov 11. PMID 27938853
- [Derived] Juraschek SP, Gelber AC, Choi HK, Appel LJ, Miller ER 3rd. Effects of the Dietary Approaches to Stop Hypertension (DASH) Diet and Sodium Intake on Serum Uric Acid. Arthritis Rheumatol. 2016 Dec;68(12):3002-3009. doi: 10.1002/art.39813. PMID 27523583
- [Derived] Amer M, Woodward M, Appel LJ. Effects of dietary sodium and the DASH diet on the occurrence of headaches: results from randomised multicentre DASH-Sodium clinical trial. BMJ Open. 2014 Dec 11;4(12):e006671. doi: 10.1136/bmjopen-2014-006671. PMID 25500372
- [Derived] Sun B, Williams JS, Svetkey LP, Kolatkar NS, Conlin PR. Beta2-adrenergic receptor genotype affects the renin-angiotensin-aldosterone system response to the Dietary Approaches to Stop Hypertension (DASH) dietary pattern. Am J Clin Nutr. 2010 Aug;92(2):444-9. doi: 10.3945/ajcn.2009.28924. Epub 2010 Jun 2. PMID 20519561
- See also: Related Info — http://www.brighamandwomens.org/patient/patient_dept_frame.asp?id=8